CLINICAL TRIAL: NCT01952925
Title: Combined Atrial Fibrillation Ablation and Renal Artery Denervation for the Maintenance of Sinus Rhythm and Management of Resistant Hypertension
Brief Title: Combined Afib Ablation and RA Denervation for the Maintenance of Sinus Rhythm and Management of Resistant Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to obtain IRB approval
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Charles Henrikson, MD, Associate Professor, Knight Cardiovascular Institute, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-D-9699
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Afib; Hypertension
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined afib ablation and RA denervation (Experimental): Patients with atrial fibrillation and resistant hypertension will be enrolled and undergo a single procedure consisting of pulmonary vein isolation and renal artery denervation.
  Interventions: Procedure: Renal Artery denervation

INTERVENTIONS:
Procedure: Renal Artery denervation — RA denervation performed as part of afib ablation procedure

SUMMARY:
The purpose of this study is to perform renal artery denervation at the same time as atrial fibrillation ablation. RA denervation may reduce blood pressure, increase the chances of a successful atrial fibrillation ablation, and decrease the number of medications required to control blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients scheduled for afib ablation
* Patient taking one or more BP medication

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
change in systolic blood pressure when measured at routine 1 and 3 month follow up appointments | 1 to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Henrikson, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States